CLINICAL TRIAL: NCT00544804
Title: A Phase I Dose Escalation Study of 5-Day Intermittent Oral Lapatinib Therapy With Biomarker Analysis in Patients With HER2-Overexpressing Breast Cancer
Brief Title: Lapatinib in Treating Patients With Advanced or Metastatic Breast Cancer That Overexpresses HER2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSF-077518
Record Dates: First submitted 2007-10-13; First posted 2007-10-16 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-07

CONDITIONS: Breast Cancer; Metastatic Cancer
Keywords: recurrent breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; bone metastases
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Lapatinib; Gene Expression Profiling

ARMS (1):
- Lapatinib (Experimental): Dose Escalation Study of 5-Day Intermittent Oral Lapatinib Therapy With Biomarker Analysis in Patients With HER2-Overexpressing Breast Cancer
  Interventions: Drug: lapatinib ditosylate; Genetic: gene expression analysis; Other: diagnostic laboratory biomarker analysis

INTERVENTIONS:
Drug: lapatinib ditosylate
Genetic: gene expression analysis
Other: diagnostic laboratory biomarker analysis

SUMMARY:
RATIONALE: Lapatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase I trial is studying the side effects and best dose of lapatinib in treating patients with advanced or metastatic breast cancer that overexpresses HER2.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose (MTD) of high-dose lapatinib ditosylate in patients with HER2-overexpressing advanced or metastatic breast cancer.
* To determine the dose-limiting toxicity of this drug in these patients.

Secondary

* To determine whether tumor HER2 can be completely inactivated by lapatinib ditosylate at its MTD in the 5-day schedule.
* To determine whether the total inactivation of HER2 decreases cardiac ejection fraction.

OUTLINE: Patients are stratified according to dose level.

Patients receive escalating doses of oral lapatinib ditosylate twice daily on days 1-5 until the maximum tolerated dose is determined. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity.

Some patients undergo tumor tissue and blood sample collection periodically for biological and correlative studies. Samples are analyzed for evidence of cardiac injury, tumor target lysis effects, and to determine if the lapatinib serum levels result in the inactivation of tumor HER2 and HER3 kinase and oncogenic signaling.

After completion of study treatment, patients are followed every 2 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Advanced or metastatic disease
  * No effective curative therapy available
* Bone-only disease allowed
* Tumor HER2 overexpression

  * HER2 3+ expression by immunohistochemistry OR > 2-fold (HER2 2+) gene amplification by fluorescence in situ hybridization
* Evaluable disease

  * Measurable disease is not required
* No progressive brain metastases
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status 0-2
* Life expectancy > 3 months
* Female
* Menopausal status not specified
* Absolute neutrophil count ≥ 1,000 cells/mm^3
* Hemoglobin ≥ 9 g/dL
* Platelet count ≥ 75,000 cells/mm^3
* Total bilirubin normal
* AST and ALT ≤ 3 x upper limits of normal (ULN) (≤ 5 x ULN with liver metastases)
* Creatinine normal OR creatinine clearance ≥ 40 mL/min
* INR ≤ 1.5
* Potassium normal
* Magnesium normal
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception prior to and during study therapy
* Cardiac ejection fraction ≥ 50%
* Consents to 2 tumor fine needle aspiration biopsies for biomarker analysis

  * Lung-only disease or sites otherwise deemed high-risk for biopsy, the requirement for biopsy will be waived

Exclusion criteria:

* History of significant cardiac disease including any of the following:

  * Congestive heart failure
  * Symptomatic cardiac arrhythmias
  * Unstable angina
* Uncontrolled prior lapatinib ditosylate therapy toxicity ≥ grade 2
* Allergic reactions to IV contrast dye despite standard prophylaxis
* History of malabsorption syndrome or disease significantly affecting gastrointestinal function or major resection of the stomach or small bowel that could affect absorption, distribution, metabolism, or excretion of study drug
* Conditions that would impair the patient's ability to swallow and retain oral medication
* Concurrent disease or condition that would make the patient inappropriate for study participation or would interfere with the patient's safety
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol

PRIOR CONCURRENT THERAPY:

* Prior lapatinib ditosylate or trastuzumab allowed
* At least 4 weeks since prior and no concurrent chemotherapy or investigational anticancer agents
* At least 2 weeks since prior and no concurrent hormonal therapy
* At least 2 weeks since prior and no concurrent lapatinib ditosylate prohibited medications, including CYP3A4 inhibitors or inducers, all herbal supplements, and gastric pH modifiers
* More than 4 weeks since prior radiotherapy
* No aspirin or plavix therapy within 7 days prior to tumor biopsy
* No concurrent coumadin

  * Low molecular weight heparin allowed provided it can be held at least 24 hours prior to tumor biopsy
* Concurrent gonadal suppression agents (i.e., Zoladex or Lupron) or palliative bisphosphonates (i.e., Zometa) allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-08; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of Lapatinib | estimated to be 12 months
  Dose Escalation of 5-Day Intermittent Oral Lapatinib Therapy With Biomarker Analysis in Patients With HER2-Overexpressing Breast Cancer

CONTACTS AND LOCATIONS:
Overall Officials: Mark M. Moasser, MD, Study Chair — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States

REFERENCES:
- [Result] Chien AJ, Munster PN, Melisko ME, Rugo HS, Park JW, Goga A, Auerback G, Khanafshar E, Ordovas K, Koch KM, Moasser MM. Phase I dose-escalation study of 5-day intermittent oral lapatinib therapy in patients with human epidermal growth factor receptor 2-overexpressing breast cancer. J Clin Oncol. 2014 May 10;32(14):1472-9. doi: 10.1200/JCO.2013.52.1161. Epub 2014 Apr 7. PMID 24711549